CLINICAL TRIAL: NCT00242801
Title: A Double Blind,Placebo Controlled,Parallel Group,Multicentre,Randomised,Phase Iii Survival Study Comparing ZD1839 (IRESSA™)(250mg Tablet) Plus Best Supportive Care Versus Placebo Plus Best Supportive Care In Patients With Advanced NSCLC Who Have Received One Or Two Prior Chemotherapy Regimens And Are Refractory Or Intolerant To Their Most Recent Regimen
Brief Title: Iressa vs Best Supportive Care - 2nd/3rd Line Survival Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1839IL/0709; ISEL
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: NSCLC
MeSH Terms: interventions — Gefitinib

INTERVENTIONS:
Drug: Gefitinib

SUMMARY:
This study is being carried out to see if adding ZD1839 to other standard supportive care is more effective than standard supportive care alone for the treatment of patients with NSCLC whose disease has recurred after previous chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* · Life expectancy of at least 8 weeks.

  * Histologically or cytologically confirmed non-small cell bronchogenic carcinoma: adenocarcinoma (including bronchoalveolar), squamous cell carcinoma, large cell carcinoma or mixed (adenocarcinoma and squamous) or undifferentiated carcinoma
  * Not suitable for chemotherapy
  * WHO Performance status 0,1, 2 or 3

Exclusion Criteria:

* Newly diagnosed CNS mets
* Less than 1 week since completion of prior radiotherapy or persistence of any radiotherapy related toxicity
* ALT/AST greater than 5 x upper limit of normal
* ANC less than 1.0 x 109/L or platelets less than 100 x 109/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1692
Dates: Start 2003-07; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to compare overall survival for ZD1839 plus best supportive care versus placebo plus best supportive care

SECONDARY OUTCOMES:
· ZD1839 + BSC versus Placebo + BSC in terms of time to treatment failure
· ZD1839 + BSC versus Placebo + BSC in terms of investigator assessed overall
· objective tumour response (CR + PR)
· ZD1839 + BSC versus Placebo + BSC in terms of tolerability
· ZD1839 + BSC versus Placebo + BSC in terms of quality of life changes

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Oncology Medical Science Direction, Study Director — AstraZeneca
Locations (211):
- Argentina (7):
  - Research Site, Capital Federal, Buenos Aires
  - Research Site, Bahía Blanca
  - Research Site, Buenos Aires
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Rosario
  - Research Site, Santa Fe
- Australia (12):
  - Research Site, Concord, New South Wales
  - Research Site, Potts Point, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Chermside, Queensland
  - Research Site, South Brisbane, Queensland
  - Research Site, Ashford, South Australia
  - Research Site, Woodville, South Australia
  - Research Site, Melbourne, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Prahran, Victoria
  - Research Site, Wodonga, Victoria
  - Research Site, Woodville South
- Brazil (6):
  - Research Site, Fortaleza, Ceará
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, São Paulo, São Paulo
  - Research Site, Sorocaba, São Paulo
- Bulgaria (6):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
- Canada (12):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Monoton, New Brunswick
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Saint Catherines, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, York, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Ste-Foy, Quebec
- Research Site, Various Cities, Chile
- Estonia (2):
  - Research Site, Talinn
  - Research Site, Tartu
- Germany (14):
  - Research Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Research Site, Heidelberg, Baden-Wurttemberg
  - Research Site, Muchen, Bavaria
  - Research Site, Frankfurt am Main, Hesse
  - Research Site, Münster, North Rhine-Westphalia
  - Research Site, Bad Segeberg, Schleswig-Holstein
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Grobhansdorf
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Hemer
  - Research Site, Mutzschen
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Marousi
  - Research Site, Thessaloniki
- Hungary (12):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Deszk
  - Research Site, Kecskemét
  - Research Site, Mosdós
  - Research Site, Mosonmagyaróvár
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Törökbálint
  - Research Site, Ujronafj
  - Research Site, Zalaegerszeg
  - Research Site, Zalaegerszeg-Pozva
- India (4):
  - Research Site, India
  - Research Site, Karnataka
  - Research Site, Kolkata
  - Research Site, Vellore
- Ireland (5):
  - Research Site, Cork, Cork
  - Research Site, Dooradoyle, Limerick
  - Research Site, Beaumont Road
  - Research Site, Dublin
  - Research Site, Elm Park
- Latvia (3):
  - Research Site, Daugavpils
  - Research Site, Liepāja
  - Research Site, Riga
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Malaysia (3):
  - Research Site, George Town
  - Research Site, Kampung Baharu Nilai
  - Research Site, Kuala Lumpur
- Mexico (9):
  - Research Site, Torreón, Coahuila
  - Research Site, Durango, Durango
  - Research Site, Guadalajara, Jalisco
  - Research Site, Monterrey, Neuvo Leon
  - Research Site, Mérida, Yucatán
  - Research Site, Acapulco
  - Research Site, Guadalajara
  - Research Site, León
  - Research Site, México
- Netherlands (7):
  - Research Site, Alkmaar
  - Research Site, Amsterdam
  - Research Site, Enschede
  - Research Site, Groningen
  - Research Site, Leiden
  - Research Site, Nieuwegein
  - Research Site, Rotterdam
- Norway (12):
  - Research Site, Ålesund
  - Research Site, Bergen
  - Research Site, Gjettum
  - Research Site, Hamar
  - Research Site, Haugesund
  - Research Site, Kristiansand
  - Research Site, Nordbyhagen
  - Research Site, Oslo
  - Research Site, Skien
  - Research Site, Stavanger
  - Research Site, Tromsø
  - Research Site, Trondheim
- Research Site, Various Cities, Peru
- Philippines (3):
  - Research Site, Manila
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (7):
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Zabrze
- Romania (5):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Timișoara
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Research Site, Singapore, Singapore
- Slovakia (13):
  - Research Site, Bratislava
  - Research Site, Dolný Kubín
  - Research Site, Kojice
  - Research Site, Martin
  - Research Site, Michalovce
  - Research Site, Nitra
  - Research Site, Nitra-Zobor
  - Research Site, Nové Zámky
  - Research Site, Poprad
  - Research Site, Poprad - Kvetnica
  - Research Site, Prejov
  - Research Site, Trnava
  - Research Site, Žilina
- Sweden (9):
  - Research Site, Västerås, Västmanland County
  - Research Site, Gothenburg
  - Research Site, Huddinge
  - Research Site, Jönköping
  - Research Site, Karlstad
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Uppsala
- Taiwan (6):
  - Research Site, Banqiao District, Taipei
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
- Research Site, Various Cities, Ukraine
- United Kingdom (36):
  - Research Site, Cambridge, Cambrideshire
  - Research Site, Exeter, Devon
  - Research Site, Colchester, Essex
  - Research Site, Romford, Essex
  - Research Site, Gorleston-on-Sea, Great Yarmouth
  - Research Site, Fulwood, Lanc
  - Research Site, Norwich, Norfolk
  - Research Site, Nottingham, Northamptonshire
  - Research Site, Belfast, Northern Ireland
  - Research Site, Birmingham, West Midlands
  - Research Site, Aberdeen
  - Research Site, Birmingham
  - Research Site, Bradford
  - Research Site, Brighton
  - Research Site, Coventry
  - Research Site, Dundee
  - Research Site, Essex
  - Research Site, Glasgow
  - Research Site, Guildford
  - Research Site, Gwynedd
  - Research Site, Harrogate
  - Research Site, Huddersfield
  - Research Site, Hull
  - Research Site, Lancaster
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Nottingham
  - Research Site, Oxford
  - Research Site, Reading
  - Research Site, Southampton
  - Research Site, Swansea
  - Research Site, Wolverhampton
  - Research Site, York
- Research Site, Various Cities, Venezuela